CLINICAL TRIAL: NCT06850870
Title: Onward Door-Through-Door Companion Rideshare Technology to Improve Care for Older Adults and Individuals With Alzheimer's Disease and Related Dementias (AD/ADRD)
Brief Title: Door-Through-Door Companion Rideshare Technology for Individuals With Alzheimer's Disease and Related Dementias (AD/ADRD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Onward Health, Inc (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OnwardRCT-2024-01 v2.0; 1R44AG085945-01A1 (NIH)
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease or Associated Disorder; Dementia; Cognitive Decline
Keywords: Transportation
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Door-through-Door Rides (Experimental): Intervention Group (D2D): Door-to-Door rideshare services with a trained companion driver.
  Interventions: Other: Door-through-door companion rideshare
- Control Group (C2C): Curb-to-Curb Rides (Active Comparator): Control Group (C2C): Standard Curb-to-Curb rideshare services.
  Interventions: Other: Curb-to-curb rideshare services

INTERVENTIONS:
Other: Door-through-door companion rideshare — Door-through-Door Companion Drivers, unlike traditional rideshare services, are certified in CPR and first aid, and undergo onboard training to support older adults, individuals with mobility impairments, and those with AD/ADRD. They are trained to observe behaviors of AD/ADRD patients, monitor and detect risk of falls, elopement, and other events that may require extra assistance or emergency care during transport. Drivers accompany riders continuously until they can hand off riders to clinicians or other caregivers, or return them to their home. Technology features in the rideshare platform enable continuity of care, for consistent rider-driver matching and matching of riders to drivers based on support needs.
  Arms: Intervention Group: Door-through-Door Rides
Other: Curb-to-curb rideshare services — Curb to curb rideshare services provided by a transportation network company (TNC) with drivers who don't have specialized training in supporting healthcare riders and who don't undergo fingerprint background checks or drug and alcohol testing.
  Arms: Control Group (C2C): Curb-to-Curb Rides

SUMMARY:
The goal of this pilot randomized controlled trial is to assess the impact of D2D rideshare services with a trained companion driver on the rate of medical appointments for older adults and individuals with AD/ADRD. Participants will be assigned either door-through-door (D2D) rideshare or curb-to-curb (C2C) rideshare services. he main question it aims to answer is:

Do D2D rideshare services reduce missed medical appointment rates compared to C2C rideshare services?

DETAILED DESCRIPTION:
A pilot randomized controlled trial (Stage 1). By stratifying on levels of cognitive impairment, i.e., no cognitive impairment vs. have mild to moderate cognitive impairment/MCI or subjective cognitive decline/SCD, the research team will randomly assign 120 riders, who have scheduled medical appointments at partner practices of Onward, to one of two groups: Onward D2D service (intervention) vs. C2C rideshare (control).

Intervention Group (D2D): Door-to-Door rideshare services with a trained companion driver.

Control Group (C2C): Standard Curb-to-Curb rideshare services.

ELIGIBILITY:
Inclusion Criteria:

* All participants (or their surrogate) have the capacity to agree to allow Onward service for transportation;
* have scheduled medical appointments at partner practices of Onward;
* ages 60+
* community-dwelling;
* 60 participants who self-reported cognitive problems, such as memory issue, or have mild cognitive impairment, subjective cognitive decline, or AD/ADRD diagnosis
* Resides and attends appointments in the following San Francisco Bay Area Counties (San Francisco, Alameda, Contra Costa, Marin, San Mateo, Sonoma)

Exclusion Criteria:

* current enrollment in another transportation study;
* already using any type of free or heavily subsized transportation service;
* enrollees with comfort care only;
* Not wheelchair bound, e.g. if using a wheelchair must be foldable and must be able to transfer
* Transient, lacking consistent long term housing
* Resides outside of the San Francisco Bay Area

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Appointment Adherence | 9 Months
  The rate of missed medical appointments (No shows and same day cancellations).

SECONDARY OUTCOMES:
Quality of Life (QOL) | 9 months
  The impact of the intervention on participants' quality of life (QOL), as measured every 3 months during the study period using the ICECAP-A (ICEpop CAPability measure for Adults) Wellbeing and Quality of Life scale.
  ICECAP-A has the following five attributes, each of which can take one of four levels ranging from full capability to no capability, higher scores are better outcomes:
  * Stability (being able to feel settled and secure)
  * Attachment (being able to have love, friendship and support)
  * Autonomy (being able to be independent)
  * Achievement (being able to achieve and progress)
  * Enjoyment (being able to have enjoyment and pleasure)
Ride Acceptance Rates | 9 Months
  Participant acceptance of the ride offered.
Ride Completion Rates | 9 Months
  The completion rate of rides scheduled, as measured by the number of ride "No Shows" relative to rides booked.
Ride Satisfaction | 9 Months
  Rider satisfaction with the rides received as rated on a 5 point star scale with 1 star being the lowest rating and 5 stars being the highest.
Transportation as a SDoH | 9 Months
  Self reported unmet transportation needs as measured via surveys conducted every 3 months during the study period using Protocol for Responding to & Assessing Patients' Assets, Risks & Experiences (PRAPARE®) SDoH questionnaire transportation questions below.
  In the past 12 months, has lack of reliable transportation kept you from medical appointments, meetings, work or from getting things needed for daily living? Yes No
  Do you have trouble finding or paying for transportation? Yes No
  Has the inability to get your medications or get to appointments for care ever resulted in an emergency room visit or required hospitalization? Yes No
Caregiver Burnout | 9 Months
  Participant caregiver ratings of caregiver burnout as measured by a survey conducted every 3 months during the study period using the HealthinAging.org Caregiver Self Assessment. Source: HealthinAging.org - https://www.healthinaging.org/tools-and-tips/caregiver-self-assessment-questionnaire
  The assessment asks 18 questions, 16 are Yes/No with scores over 10 "Yes" indicating burnout, and 2 on a 1-10 scale with scores over 6 indicating burnout.
Rider Loneliness and Social Isolation | 9 Months
  Loneliness and Social Isolation will be measured every 3 months using the UCLA 3-Item Loneliness Scale.
  1. First, how often do you feel that you lack companionship: Hardly ever (1), some of the time (2), or often (3)?
  2. How often do you feel left out: Hardly ever (1), some of the time (2), or often (3)?
  3. How often do you feel isolated from others: Hardly ever (1), some of the time (2), or often (3)?
  Scoring: Sum the total of all items. Higher scores indicate greater degrees of loneliness. Possible range of scores from 3 to 9. Researchers in the past have grouped people who score 3 - 5 as "not lonely" and people with the score 6 - 9 as "lonely".

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Wachter Petty, MBA, Principal Investigator — Onward Health, Inc
Locations (1):
- Onward Health HQ, San Leandro, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: The Individual Participant Data (IPD) and supporting information will be made available starting 12 months after the completion of the study's primary endpoint analysis. Data will remain accessible for a period of 5 years following the final study report submission to ensure availability for secondary research and validation purposes.
Access Criteria: Qualified researchers and institutions engaged in health disparities, transportation accessibility, and aging-related research will be able to access individual participant data (IPD) and supporting information. Access will be granted to de-identified data to ensure participant confidentiality.
  Approved users will be able to access the following:
  De-identified Individual Participant Data (IPD) Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)
  Researchers will be required to submit a data access request, including a brief research proposal and data use agreement (DUA), outlining how the data will be used. Access will be provided through a secure data repository upon approval.